CLINICAL TRIAL: NCT01987128
Title: Blocco Del Nervo Sciatico al Poplite, Intraneurale o Extraneurale? Confronto Prospettico, Randomizzato in Cieco Tra la modalità di Iniezione di Anestetico Locale Per il Blocco Eco Guidato Del Nervo Sciatico al Poplite Nella Chirurgia Dell'Alluce Valgo
Brief Title: Popliteal Sciatic Nerve Block: Intraneural or Extraneural?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, Medical Doctor, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOGPGC04-13
Record Dates: First submitted 2013-11-05; First posted 2013-11-19 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus | interventions — Ropivacaine; Needles

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intraneural injection (Experimental): All patients in the arm will receive a single intraneural injection of 12 ml Ropivacaine 1% BBraun, Germany, in the sciatic nerve under echographic guidance.
  Interventions: Procedure: Intraneural injection; Drug: Ropivacaine; Device: PAJUNK SonoPlex 22G needle.
- extraneural injection (Active Comparator): All patients in the arm will receive a single extraneural injection of 12 ml Ropivacaine 1% BBraun, Germany, around the sciatic nerve under echographic guidance.
  Interventions: Procedure: Extraneural injection; Drug: Ropivacaine; Device: PAJUNK SonoPlex 22G needle.

INTERVENTIONS:
Procedure: Intraneural injection — BBraun Ropivacaine 1% 12ml injection divided in each sciatic components under echographic guidance with a PAJUNK SonoPlex 22G needle.
  Arms: Intraneural injection
Procedure: Extraneural injection — BBraun Ropivacaine 1% 12ml extraneural injection around sciatic nerve under echographic guidance with a PAJUNK SonoPlex 22G needle.
  Arms: extraneural injection
Drug: Ropivacaine
Device: PAJUNK SonoPlex 22G needle.

SUMMARY:
Aim of this study is to demonstrate the advantages of intraneural injection over extraneural injection in terms of onset and duration on peripheral block. In addition we will evaluate the frequency of possible adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II

Exclusion Criteria:

* Neurological diseases
* Diabetes
* Allergies to used drugs
* Chronic pain in treatment
* Electrophysiological alterations at time zero analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
onset time | every 2 minutes for a maximum of 30 minutes
  Pinprick test evaluation on sciatic nerve territory:
  With a 22G needle the blinded operator will assess sensitiveness to puncture and then assign a score every 2 minutes for 30 minutes. A score of 0 will describe no sensation to puncture, on the other hand a score of 1 will be assigned if sensation to puncture is still present.
  Evaluation of motor blockade:
  Plantar and dorsal flexion of the foot will be evaluated for motor blockade of sciatic nerve. A score of 1 will be assigned if foot movement is conserved, 2 if is impaired and 3 when disappears.
  Onset time is described as the time at which pinprick score turns to 0 and motor blockade score turns to 3.

SECONDARY OUTCOMES:
success rate in each group | at 30 minutes
  Success rate is described as the percentage of subjects with an onset time within 30 minutes in a group among all subjects treated in that group
Nerve injuries | 1, 5 weeks and at 6 months after surgery
  Neurophysiological and clinic evaluation will be assessed either with clinical examination and electrophysiological tests by a neurophysiologist eventually evidencing any movement impairment or dysesthesia in the sciatic territory.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Cappelleri, MD, Principal Investigator — ASST Gaetano Pini-CTO
Locations (1):
- Istituto Ortopedico G. Pini, Milan, Milano, Italy

REFERENCES:
- [Derived] Cappelleri G, Cedrati VL, Fedele LL, Gemma M, Camici L, Loiero M, Gallazzi MB, Cornaggia G. Effects of the Intraneural and Subparaneural Ultrasound-Guided Popliteal Sciatic Nerve Block: A Prospective, Randomized, Double-Blind Clinical and Electrophysiological Comparison. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):430-7. doi: 10.1097/AAP.0000000000000413. PMID 27281720